CLINICAL TRIAL: NCT05788848
Title: Virtual Reality Cognitive Therapy for Alzheimer's Disease
Acronym: VRCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Claritytek, Inc. (Industry)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A21-230; R43AG076169 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This study is a phase I, feasibility study for research and development of a product. We will use a single group, pre-post study design.
Who Masked: Participant
Masking Description: This study is a phase I, feasibility study for research and development of a product. We will use a single group, pre-post study design. Individuals with mild to moderate CI (diagnosis of mild cognitive impairment (MCI), probable Alzheimer's disease (AD), or Alzheimer's disease Related Dementias (ADRD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: VRCT — The VRCT will focus primarily on skills that impact instrumental activities of daily living (e.g., taking medications, shopping). Thirty-six individuals with mild to moderate AD/ADRD will be enrolled and will utilize the VRCT over seven weeks within their home.

SUMMARY:
To evaluate the usability, feasibility, and acceptability of VRCT iteratively on 36 AD/ADRD individuals with mild to moderate CI.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) and Alzheimer's disease-related Dementias (ADRD) resulting in cognitive decline affects more than 5.8 million Americans. Given the impact on quality of life, there is a great need for therapies focused on cognition. In this study, we will test the feasibility, usability, and acceptability of a novel Virtual Reality Cognitive Therapy (VRCT) for AD developed by ClarityTek, Inc. The VRCT will focus primarily on skills that impact instrumental activities of daily living (e.g., taking medications, shopping). Thirty-six individuals with mild to moderate AD/ADRD will be enrolled and will utilize the VRCT over seven weeks within their home. Enrollment will occur in cohorts of 12 individuals, so that the VRCT can be revised and optimized based on the results, prior to the next cohort. We will also hold Expert Focus Groups with clinician specialists to obtain feedback for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild cognitive impairment (MCI), probable Alzheimer's disease (AD) or Alzheimer's disease Related Dementias (ADRD)
* Montreal Cognitive Assessment (MoCA) score of 11-25
* Age 30-89

Exclusion Criteria:

* Non-English speaking
* History of seizure disorder, vertigo disorder, or severe motion sickness that would impact their ability to participate in the intervention
* History of any other serious condition that may limit their ability to participate in the intervention, as determined by the investigators.
* Inability to use the VR device (e.g., severe visual/hearing impairment, aphasia, facial injuries)

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and Usability of Virtual Reality Cognitive Therapy (VRCT) for Alzheimer's Patients: Assessment of Patient-Reported Simulator Sickness and System Usability using The Simulator Sickness Questionnaire and System Usability Scale | from baseline at 7 weeks
  Patient-Reported Simulator Sickness and System Usability using The Simulator Sickness Questionnaire and System Usability Scale Questionnaire
Acceptability of Virtual Reality Cognitive Training (VRCT) for Alzheimer's Patients: Assessment of Patient-Reported Acceptability using Free-Form Suggestion Feedback | from baseline at 7 weeks
  Patient-reported Acceptability of VRCT using Free-Form Suggestion Feedback such as acceptable, not acceptable or acceptable with changes.

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living (IADL) performance | from baseline at 7 weeks
  The IADL performance measured by change in The Lawton IADL performance
Cognitive Impairment (CI) | from baseline at 7 weeks
  Cognitive Impairment measured by change in the Cognitive Failures Questionnaire (CFQ)
Anxiety and Depression | from baseline at 7 weeks
  Anxiety and Depression will also be measured by change in the Hospital Anxiety-Depression Scale (HADS) to monitor as a potential confounder of cognition and function.

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Hanson, PhD, Principal Investigator — HealthPartners Neuroscience Center
Locations (1):
- HealthPartners, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided